CLINICAL TRIAL: NCT06983431
Title: DIGITALIZATION OF PERSONALISED HEALTH RISK MANAGEMENT IN AT-RISK GROUPS TO IMPROVE HEALTH OUTCOMES THROUGH INTEGRATION OF TECHNOLOGICAL AND SOCIAL INNOVATION
Brief Title: DIGITALIZATION OF PERSONALISED HEALTH RISK MANAGEMENT
Acronym: DIG4HEALTH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Slovak Academy of Sciences (Other Government)
Collaborators: University Hospital Bratislava Comenius University (Unknown); Kempelen Institute of Inteligent Technologies (Unknown)
Responsible Party: Principal Investigator, Jozef Ukropec, PhD, DSc, Slovak Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 09I05-03-V02-00060
Record Dates: First submitted 2025-04-29; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-04

CONDITIONS: Pre-obesity; Obesity
Keywords: wearable; behavioural intervention; habitual physical activity; quality of life; body weight and composition; sleep duration / eficiency; heart rate variability
MeSH Terms: conditions — Obesity; Body Weight

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into one of the four intervention groups:
  1. Self coaching (technology-assisted online intervention)
  2. Health coaching - online contact with professional coach
  3. Peer coaching - online contact with peer-coach
  4. Control group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Self coaching (technology-assisted online intervention) (Experimental): Self coaching (technology-assisted online intervention)
  Interventions: Behavioral: technology driven self coaching
- Health coaching - online contact with professional coach (Experimental): Health coaching - online contact with professional coach
  Interventions: Behavioral: Health coaching
- Peer coaching - online contact with peer-coach (Experimental): Peer coaching - online contact with peer-coach
  Interventions: Behavioral: Peer coaching
- Control group. (Active Comparator): Wearable and basic information on healthy lifestyle will be provided, but any of the coaching strategies will be applied
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: technology driven self coaching — subject will be provided with the technology driven lifestyle coaching based on the real time data from the wearables
  Arms: Self coaching (technology-assisted online intervention)
Behavioral: Health coaching — participants will be provided with the health coach (expert) driven lifestyle coaching based on the real-time data from the wearables
  Arms: Health coaching - online contact with professional coach
Behavioral: Peer coaching — participants will be provided with the peer coach (expert) driven lifestyle coaching based on the real-time data from the wearables
  Arms: Peer coaching - online contact with peer-coach
Behavioral: Active Control — participants will be provided with the wearable, but not exposed to any of the coaching strategies. Real-time data provided by the wearable will be available to them.
  Arms: Control group.

SUMMARY:
The principal objective of the project is:

* to bring together academic and business research organisations in a joint partnership integrating technological and social innovation,
* in order to develop proof-of-concept of a scalable and cost effective personalised digital health program for (pre)obesity patients,
* by integrating, in an ethical manner, adaptive AI components aimed at personalisation of the program as well as its cost management,
* with the ultimate objective to support sustained behavioural change leading to adoption and internalisation of healthy lifestyle choices.

DETAILED DESCRIPTION:
This research project is aimed at leveraging digital tools to personalise preventive healthcare interventions for at-risk populations in ways that address the above-mentioned challenges. At risk populations, in the context of this project, generally means: Younger to middle aged (aged 30-50) sedentary individuals with (pre)obesity expressing behavioural, clinical, biochemical and anamnestic indicators of increased risk for accelerated decline of cardio-metabolic and cognitive health.

Primary outcomes will be the rate of wearable adoption/use, individualised behavioural change persistence and elicited health benefit

Secondary outcomes will include step count, activity of medium & vigorous intensity, sleep duration/efficiency, heart rate, quality of life, body weight, body composition, blood pressure, and level of fitness as determined by the wearable or validated questionaires available on the landing page.

Participants will be randomly assigned into one of the three intervention groups and a control group. The three intervention groups:

1. Self-health coaching will be conducted using wearable and technology provided nudges allowing personalised technology-assisted real-time feedback. With this approach, on-line intervention with minimal human resource costs and high technology involvement with a potential to deliver sustainable and cost-effective behavioural change to a large at-risk population will be tested.

   This intervention approx. 80 participants will be examined for the duration of 14 weeks. Long term follow up examination is envisaged, but it is beyond this study duration and will be supported by subsequent funding.
2. Health coaching (online health-coach community based) intervention will be based on applying wearable providing the most effective impact on health-related outcomes as evidenced in the exploratory study in combination with the online supervised intervention by the professional health-coach in an online group (community setting). Within this intervention the efficacy of an online supervised health coaching applied in community settings will be tested. Professional health coaching strategy using wearable-related outcomes will be provided as a golden standard of the behavioural intervention with proven efficiency. This intervention will be tested on approx. 80 participants for the duration of 14 weeks.
3. Peer coaching: Peers will be identified from the study population based on their response to specific community challenges. Natural leader characteristics will be deciphered from knowledge provided by the past supervised community-based behavioural interventions at BMC SAS and the other open sources subjected to AI driven prediction modelling. Within this intervention the efficacy of an online health coaching led by peers will be tested in an online community based setting. Peer-based health coach will lead participants through health training based on the "protocol" defining minimal coaching criteria but imposing no limits to any communication activities including the real-time access to the wearable-provided outcomes. The intervention will be tested on approx. 80 participants for the duration of 14 weeks. Long term follow up examination is envisaged, but it is beyond this study duration and will be supported by subsequent funding.
4. Control group participants will receive health coaching - related information enabling self-health coaching in a printed form during initial phenotyping visit and a wearable. The control group will consist of approx. 50 participants and observation period will be 14 weeks. Long term follow up examination is envisaged, but it is beyond this study duration and will be supported by subsequent funding.

Innovative strategies to employ AI and machine learning will be tested to support their meaningful (providing real health benefits) and cost effective use.

ELIGIBILITY:
Inclusion Criteria:

* obesity (BMI 27-42 kg/m²)
* capacity and willingness to use smartphone
* capacity and willingness to use wearables
* readiness to change (validated questionaire)

Exclusion Criteria:

* diseases that prevent participation in the program, or insufficiently controlled diseases, or terminal-stage illnesses
* excessive alcohol consumption or a history of other addictions
* patients currently participating in a weight-loss program (commercial, medically supervised, or a research study)
* patients using anti-obesity medications who are in the dosage adjustment phase within the last four weeks
* patients who are not mentally, physically, or technologically capable of participating
* patients who are unable to provide informed consent
* patients not adhering to the study protocol

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of wearable adoption/use | 24 months
  Rate of wearable adoption/use will be determenrd from the wearable allowed data in-flow.
Effect of intervention on Quality of life | 24 months
  Quality of life will be provided by the validated questionaire filled in at baseline and after completing the study.
Effect of intervention on health | 24 months
  Effects of intervention for health state will be provided by the questionaire administered at the baseline and after completing the study.

SECONDARY OUTCOMES:
Habitual physical activity volume | 24 months
  wearable (Garmin vivosmart 5) provided daily step count
Sleep quality | 24 months
  wearable (Garmin vivosmart 5) provided sleep quality parameter
Activity-related energy expenditure | 24 months
  Wearable (Garmin - vivosmart 5) provided daily active calories measure.
Stress level | 24 months
  Wearable (GARMIN vivosmart 5) provided measure of daily stress level

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Ukropec, PhD, DSc, Principal Investigator — Biomedical Research Center Slovak Acad Sci; Zuzana Košutzka, A/prof., PhD, Study Chair — University Hospital Bratislava and Faculty of Medicine Comenius University; Emília Sičáková - Beblavá, Prof. Ing. PhD, Study Director — University Hospital Bratislava and Faculty of Medicine Comenius University; Miroslav Beblavý, A/prof. PhD, Study Director — University Hospital Bratislava and Faculty of Medicine Comenius University
Locations (1):
- Center for Obesity Management EASO, Biomedical Research Center SAS, Bratislava, Bratislava Region, Slovakia

IPD SHARING:
Plan to Share IPD: No
Data will be provided in scientiffic publications. Anz data related to this study could be available upon reasonable request after their publication.